CLINICAL TRIAL: NCT00003747
Title: Phase I (Tumour Site Specific) Study of Carboplatin and Temozolomide in Patients With Advanced Melanoma
Brief Title: Carboplatin and Temozolomide in Treating Patients With Unresectable or Metastatic Melanoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mount Vernon Cancer Centre at Mount Vernon Hospital (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066867; MTVERNHOSP-OCT1998; EU-98069
Record Dates: First submitted 1999-11-01; First posted 2004-05-21 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2001-03

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Carboplatin; Temozolomide

INTERVENTIONS:
Drug: carboplatin
Drug: temozolomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining carboplatin and temozolomide in treating patients who have unresectable or metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of carboplatin and temozolomide in patients with unresectable or metastatic melanoma. II. Assess the safety of this cytotoxic combination in this patient population. III. Assess the preliminary evidence of efficacy of this combination in these patients.

OUTLINE: This is an open label, dose escalation study. Patients receive oral temozolomide once daily on days 1-5. Carboplatin IV is administered over 1 hour on day 1. Courses are repeated every 28 days. Treatment continues for a maximum of 6 courses in the absence of toxicity and disease progression. Sequential dose escalation of carboplatin with a fixed dose of temozolomide is followed by sequential dose escalation of carboplatin at a higher fixed dose of temozolomide. Dose escalation in cohorts of 3-6 patients each continues until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose limiting toxic effects. If the combination treatment with carboplatin given on day 1 of temozolomide therapy is more toxic than anticipated, then the study is repeated with carboplatin given on day 5 of temozolomide therapy. Patients are followed at least every 2 months.

PROJECTED ACCRUAL: Approximately 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven unresectable or metastatic melanoma

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: ECOG 0-2 Life expectancy: Greater than 3 months Hematopoietic: Hemoglobin greater than 10 g/dL WBC greater than 3,000/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin less than 1.8 mg/dL AST less than 3 times upper limit of normal (ULN) Alkaline phosphatase less than 3 times ULN No hepatitis B Renal: Creatinine less than 1.4 mg/dL OR Creatinine clearance greater than 50 mL/min Cardiovascular: No New York Heart Association class II cardiac disease Pulmonary: No pulmonary disease requiring oxygen therapy Other: Not pregnant Fertile patients must use effective contraception during study and for 3 months following No concurrent serious nonmalignant disease No AIDS No uncontrolled infection No uncontrolled diabetes No medical condition that will interfere with taking oral temozolomide

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior biologic therapy and recovered No concurrent biologic therapy Chemotherapy: At least 4 weeks since prior chemotherapy and recovered No prior carboplatin and temozolomide No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy and recovered At least 3 weeks since prior palliative radiotherapy No concurrent radiotherapy Surgery: No concurrent surgery to tumor Other: No other concurrent investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1998-10

CONTACTS AND LOCATIONS:
Overall Officials: Gordon J.S. Rustin, MD, Study Chair — Mount Vernon Cancer Centre at Mount Vernon Hospital
Locations (1):
- Mount Vernon Hospital, Northwood, England, United Kingdom